CLINICAL TRIAL: NCT05993403
Title: The Effect of The Cultural Sensitivity Education Program Applied to Nurses on The Level of Intercultural Sensitivity and Compassion
Brief Title: The Cultural Sensitivity Education Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sultan Ayaz Alkaya (Other)
Responsible Party: Sponsor-Investigator, Sultan Ayaz Alkaya, Prof. Dr., Faculty of Nursing, Nursing Department, Dean of the Faculty of Nursing, Gazi University
Organization: Gazi University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2023-558520
Record Dates: First submitted 2023-08-08; First posted 2023-08-15 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2023-08

CONDITIONS: Intercultural Sensitivity
Keywords: Compassion; Intercultural sensivity; Nursing

STUDY DESIGN:
Intervention Model Description: The study was conducted with a randomized controlled experimental design to determine the effect of intercultural sensitivity training applied to nurses on intercultural sensitivity and compassion level.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intercultural Sensitivity Education (Experimental): Data collection tools were applied to this group before the research. A training program consisting of three sessions was applied to the intervention group. Each training session lasted an average of 90-100 minutes. Various methods and techniques were used in the trainings.
  Interventions: Other: Intercultural Sensitivity Education Program
- Control (No Intervention): Data collection tools were applied to this group before the research. No intervention was applied to this group.

INTERVENTIONS:
Other: Intercultural Sensitivity Education Program — The training program consists of three sessions. In the Intercultural Sensitivity training for nurses, it was aimed to develop the level of intercultural sensitivity, and it was aimed to provide proficiency in providing services to raise awareness and knowledge about intercultural sensitivity.
  Arms: Intercultural Sensitivity Education

SUMMARY:
The research was carried out with a randomized controlled experimental design in order to determine the effect of intercultural sensitivity training applied to nurses on intercultural sensitivity and compassion level. Nurses working in a private hospital were included in the sample of the study. A total of 66 nurses, 32 of whom were in the intervention and control groups, were included in the study. "Personal Information Form", "Intercultural Sensitivity Scale" and "Compassion Scale" were used to collect data. "Intercultural Sensitivity Training" consisting of four sessions was given to the intervention group.

DETAILED DESCRIPTION:
Within the scope of the research, an intercultural sensitivity training program for nurses was created. The training program was implemented and an evaluation was made after the implementation.

ELIGIBILITY:
Inclusion Criteria:

* Being a nurse working under the Nursing Services Directorate
* Volunteering to participate in research

Exclusion Criteria:

* Having a disease that prevents participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-10-21 (Actual)

PRIMARY OUTCOMES:
Intercultural Sensitivity Level (Intercultural Sensitivity Scale) | before the implementation
  The Intercultural Sensitivity scale is a five-point Likert type and consists of 24 items. The lowest total score that can be obtained from the scale was calculated as 24 and the highest score as 120. An increase in the score obtained from the scale indicates an increase in the level of intercultural sensitivity.
Intercultural Sensitivity Level (Intercultural Sensitivity Scale) | four weeks after the start of application
  The Intercultural Sensitivity scale is a five-point Likert type and consists of 24 items. The lowest total score that can be obtained from the scale was calculated as 24 and the highest score as 120. An increase in the score obtained from the scale indicates an increase in the level of intercultural sensitivity.
Intercultural Sensitivity Level (Intercultural Sensitivity Scale) | three months after the finish of implementation
  The Intercultural Sensitivity scale is a five-point Likert type and consists of 24 items. The lowest total score that can be obtained from the scale was calculated as 24 and the highest score as 120. An increase in the score obtained from the scale indicates an increase in the level of intercultural sensitivity.

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)